CLINICAL TRIAL: NCT02850341
Title: Step Away From Depression - Evaluation of a Pedometer Intervention With Inpatients With Major Depression - A Randomized Controlled Trial
Brief Title: Step Away From Depression - Evaluation of a Pedometer Intervention With Inpatients With Major Depression
Acronym: SAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Robert-Enke-Stiftung (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. Andreas Ströhle, Prof. Dr. med., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SAD
Record Dates: First submitted 2016-07-22; First posted 2016-08-01 (Estimated); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Depression
Keywords: Physical Activity; Mental Health; Health Behavior; Walking; Physical Exercise; Mental disorder
MeSH Terms: conditions — Depression; Motor Activity; Psychological Well-Being; Health Behavior; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Patients receive a pedometer and instructions how to raise their physical activity
  Interventions: Device: Pedometer
- Control group (No Intervention): Patients receive treatment-as-usual

INTERVENTIONS:
Device: Pedometer — Patients receive a pedometer with instructions how to raise their number of daily steps
  Arms: Intervention group

SUMMARY:
The purpose of this study is to determine if the use of pedometers can help depressive inpatients in psychiatric clinics to increase their level of physical activity. Therefore patients are given a pedometer and instructions how to raise their level of daily steps. Intervention group is compared with a control group that is receiving treatment-as-usual. The intervention is hypothesized to increase number of daily steps and have positive effects on mood, depression and anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Major Depression, moderate to severe as main diagnosis
* Inpatient status
* Prospected inpatient treatment of at least 4 weeks
* Able to understand german

Exclusion Criteria:

* Physical disease or disability that makes it impossible to reach the goal 5000 steps per day
* Borderline personality disorder
* Bipolar Disorder
* Schizophrenia
* Anorexia Nervosa
* Dementia
* Psychotic Depression
* Pregnancy
* Acute suicidality
* Substance dependancies with actual consumption (except nicotine)
* Current pedometer-use
* More than 10.000 steps per day

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Change in average number of steps per day | From baseline (1.-3. day of inpatient treatment) to end of inpatient treatment (3 days before end of inpatient treatment)
  Number of steps per day is objectively measured using accelerometry (ActiGraph GT1M)
Change in depressive symptoms - clinician rated | From baseline (1.-3. day of inpatient treatment) to end of inpatient treatment (3 days before end of inpatient treatment)
  Depressive symptoms are rated by a blind study employee using MADRS

SECONDARY OUTCOMES:
Change in physical activity - subjective | From baseline (1.-3. day of inpatient treatment) to end of inpatient treatment (3 days before end of inpatient treatment)
  Physical activity is subjectively measured with the International Physical Activity Questionnaire (IPAQ)
Change in physical activity - objective | From baseline (1.-3. day of inpatient treatment) to end of inpatient treatment (3 days before end of inpatient treatment)
  Physical activity is objectively measured using accelerometry (ActiGraph GT1M)
Change in psychopathological symptoms | From baseline (1.-3. day of inpatient treatment) to end of inpatient treatment (3 days before end of inpatient treatment)
  Psychopathological symptoms are measured by the Symptom Checklist 27 (SCL-27)
Change in health-related quality of life | From baseline (1.-3. day of inpatient treatment) to end of inpatient treatment (3 days before end of inpatient treatment)
  Health-related quality of life is measured using the Short-Form Health Questionnaire (SF-12)
Change in depressive symptoms | From baseline (1.-3. day of inpatient treatment) to end of inpatient treatment (3 days before end of inpatient treatment)
  Depressive symptoms are measured using the Beck Depression Inventory (BDI II)
Change in anxiety symptoms | From baseline (1.-3. day of inpatient treatment) to end of inpatient treatment (3 days before end of inpatient treatment)
  Anxiety symptoms are measured using the Beck Anxiety Inventory (BAI)
Change in self-efficacy for physical activity | From baseline (1.-3. day of inpatient treatment) to end of inpatient treatment (3 days before end of inpatient treatment)
  Self-efficacy for physical activity is measured using six likert scaled items by Scholz, U., Sniehotta, F. & Schwarzer, R. (2005)
Change in intention for physical activity | From baseline (1.-3. day of inpatient treatment) to end of inpatient treatment (3 days before end of inpatient treatment)
  Intention for physical activity is measured using two likert scaled items by Sniehotta, F. F., Schwarzer, R., Scholz, U., & Schüz, B. (2005)
Change in self concordance of the motivation for physical activity | From baseline (1.-3. day of inpatient treatment) to end of inpatient treatment (3 days before end of inpatient treatment)
  Self concordance of the Motivation for physical activity is measured using the "Sport- und bewegungsbezogene Selbstkonkordanz Skala", which consists of 12 likert scaled items
Change in outcome expectancies for physical activity | From baseline (1.-3. day of inpatient treatment) to end of inpatient treatment (3 days before end of inpatient treatment)
  Outcome expectancies for physical activity are measured using 6 likert scaled items by Lippke S., Ziegelmann, J. P. & Schwarzer, R. (2005)
Change in planning and barrier planning for physical activity | From baseline (1.-3. day of inpatient treatment) to end of inpatient treatment (3 days before end of inpatient treatment)
  Planning and barrier planning for physical activity is measured using 8 likert scaled items by Sniehotta, F. F. et al. (2005) / Renner, B. (2007)
Duration of inpatient treatment (Number of days) | Duration of inpatient treatment is assessed at the end of inpatient treatment
Change in general self-efficacy | From baseline (1.-3. day of inpatient treatment) to end of inpatient treatment (3 days before end of inpatient treatment)
  General self-efficacy is measured using the General-Self-Efficacy Scale (GSE)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Ströhle, Prof.Dr., Principal Investigator — Charité Universitätsmedizin Berlin - Klinik für Psychiatrie und Psychotherapie
Locations (9):
- Paracelsus University Salzburg - Clinic for Psychiatry and Psychotherapy, Salzburg, Austria
- Germany (8):
  - Ludwig Maximilian University Munich - Clinic for Psychiatry and Psychotherapy, Munich, Bavaria
  - Oberhavel Clinics GmbH - Clinic for Psychiatry, Psychosomatics and Psychotherapy, Hennigsdorf, Brandenburg
  - Health Center Odenwaldkreis GmbH - Center for Mental Health, Erbach im Odenwald, Hesse
  - University of Frankfurt/Main - Clinic for Psychiatry, Psychosomatic and Psychotherapy, Frankfurt am Main, Hesse
  - University of Göttingen - Clinic for Psychiatry and Psychotherapy, Göttingen, Lower Saxony
  - University RWTH Aachen, Clinic for Psychiatriy, Psychotherapy and Psychosomatic, Aachen, North Rhine-Westphalia
  - Ev.Luth. Diakonissenanstalt Flensburg - Clinic for Psychiatry, Psychosomatic and Psychotherapy, Flensburg, Schleswig-Holstein
  - Charité Universitätsmedizin Berlin - Departement of Psychiatry, Berlin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.angstambulanz-charite.de